CLINICAL TRIAL: NCT06507696
Title: Comparison of the Efficacy of Ice and Soaked Gauze in Managing Early Postoperative Thirst
Brief Title: Comparison of the Efficiency of Two Different Methods in Managing Early Postoperative Thirst
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Yasemin Uslu, Assoc. Prof., Acibadem University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-21/01
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Patient Satisfaction; Nursing Caries; Post-Op Complication
Keywords: thirst management; postoperative care; surgical patient; surgical thirsty
MeSH Terms: conditions — Patient Satisfaction; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Randomized controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ice Application (Experimental): * In ice application, 5 ml of drinking water was filled in a 10 ml syringe and frozen by inserting a plastic piston into it and then these frozen ice cubes were given into the mouths of the patients.
  * The ice cubes were prepared before the application and stored in the freezer section of the refrigerator.
  * The ice was taken out of the frozen syringe and the nurse moved it around the patient's mouth to melt it.
  * By holding the ice cubes from the piston part to the researcher, the patient was allowed to suck and melt them in the mouth.
  Interventions: Other: Ice Application
- Wetted Gauze Application (Experimental): * During wetted gauze application, sterile gauze swabs were wetted with drinking water.
  * Sterile gauze swabs (10 cm*10cm) were wetted with 5 ml and applied for 5 minutes.
  * The wetted end part of the gauze swabs was allowed to be sucked in the patient's mouth by the researcher.
  Interventions: Other: Wetted Gauze Application
- No intervention (No Intervention): Patients in the control group did not receive any application

INTERVENTIONS:
Other: Ice Application — Drinking water was placed in a syringe and filled in the refrigerator
  Arms: Ice Application
Other: Wetted Gauze Application — Sterile gauze soaked with drinking water
  Arms: Wetted Gauze Application

SUMMARY:
Postoperative thirst is one of the most common problems in patients. Thirst is a subjective symptom. Thirst can cause unwanted problems in patients such as anxiety, discomfort and nausea. It may even cause anxiety, hypertension, dysrhythmia, non-compliance with treatment and increased need for anesthesia. Although different methods have been applied in the management of thirst in the existing literature and positive results have been obtained, studies with high evidence value are very limited. The aim of this study was to compare the effectiveness of two different methods in thirst management.

DETAILED DESCRIPTION:
In this study, the investigators compared the effectiveness of two of the methods proposed in the literature for the relief of postoperative thirst.

These methods are ice application and wet gauze. A numerical comparison scale was used to assess and monitor thirst (0=no thirst, 10=worst perceived thirst).

In patients with a thirst score of 4 and above in the early postoperative period, the duration of thirst severity and the method of quenching thirst with oral ice or wet gauze impregnation were compared. In addition, a control group without any intervention was included. The thirst conditions of these three groups were compared.

A total of 240 patients, 80 in each group, were included in the study. Oral ice was applied in one group, wet gauze in the second group and no intervention was applied in the third group.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years
* undergoing elective surgery
* Patients undergoing surgery other than gastrointestinal system surgery
* Patients in class I, II, III according to the American anesthesiologists' association classification (ASA)
* Patients who have completed a minimum of 6 hours of strict fasting and 3 hours of thirst
* Patients who can verbally express a thirst level of 4 points or more according to visual benchmark scale in the early postoperative period
* Patients who comply with the safety protocol in the early postoperative period
* Patients who can express their thirst in the early postoperative period/recovery unit
* Patients with a duration of surgical anesthesia ≥1 hour and taken to the recovery unit at the end of surgery will be included in the study.

Exclusion Criteria:

* Emergency planned surgeries
* Patients who had a second surgical intervention during the hospitalization period
* Patients who need intensive care after surgery
* Patients with problems in the extubation process after surgery
* Patients with altered state of consciousness after surgery
* Patients with fluid electrolyte imbalance (hypovolemia and sodium imbalance)
* Patients with swallowing difficulties and fluid intake restriction
* Foreign patients with language barriers
* Patients with menthol allergy
* Patients with problems in the head, neck, throat and mouth will be excluded from the sample.
* Women who have just given birth and are breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Thirst score | Using Thirst Visual Comparion Scale score after immediately after surgery (T1) 5th min.(T2), 30th min.(T3), 60th min.(T4), 90th min.(T5)
  Visual Comparion Scale (VCS) was used to assess thirst. In this scale, thirst was graded from 0 to 10. 0=no thirst, 10=the most severe thirst.
  The scale was evaluated as 0-3 points mild thirst, 4-6 points moderate thirst, 7-10 points severe thirst.
  * First follow-up (T1): Patient's thirst level measured by VCS and intervention (ice application or wet gauze application)
  * Second follow-up (T2); evaluation was performed with VCS 5 minutes after the application.
  * Third follow-up (T3); evaluation was performed with VCS 30 minutes after the application.
    * Fourth follow-up (T4); assessment was performed with VCS 60 minutes after the application.
  Fifth follow-up (T5); evaluation was performed with VCS 90 minutes after the application.
  The thirst level of the patient was measured 5 times in total. At 90 minutes, data collection was terminated.
  Scores between 5 measurement values were compared.

CONTACTS AND LOCATIONS:
Overall Officials: Fevzi Toraman, Prof. Dr., Study Director — Acıbadem Mehmet Ali Aydınlar Üniversitesi
Locations (2):
- Turkey (Türkiye) (2):
  - Yasemin Uslu, Istanbul, Ataşehir
  - Acıbadem University, Istanbul, Eyalet/Yerleşke

REFERENCES:
- [Result] Serato VM, Fonseca LF, Birolim MM, Rossetto EG, Mai LD, Garcia AKA. Package of menthol measures for thirst relief: a randomized clinical study. Rev Bras Enferm. 2019 Jun 27;72(3):600-608. doi: 10.1590/0034-7167-2018-0057. English, Portuguese. PMID 31269122
- [Result] Peyrot des Gachons C, Avrillier J, Gleason M, Algarra L, Zhang S, Mura E, Nagai H, Breslin PA. Oral Cooling and Carbonation Increase the Perception of Drinking and Thirst Quenching in Thirsty Adults. PLoS One. 2016 Sep 29;11(9):e0162261. doi: 10.1371/journal.pone.0162261. eCollection 2016. PMID 27685093
- [Result] Nascimento LAD, Garcia AKA, Conchon MF, Aroni P, Pierotti I, Martins PR, Nakaya TG, Fonseca LF. Advances in the Management of Perioperative Patients' Thirst. AORN J. 2020 Feb;111(2):165-179. doi: 10.1002/aorn.12931. PMID 31997333
- [Result] Nascimento LA, Fonseca LF, Rosseto EG, Santos CB. [Development of a safety protocol for management thirst in the immediate postoperative period]. Rev Esc Enferm USP. 2014 Oct;48(5):834-43. doi: 10.1590/s0080-6234201400005000009. Portuguese. PMID 25493487
- [Result] Conchon MF, Fonseca LF. Efficacy of an Ice Popsicle on Thirst Management in the Immediate Postoperative Period: A Randomized Clinical Trial. J Perianesth Nurs. 2018 Apr;33(2):153-161. doi: 10.1016/j.jopan.2016.03.009. Epub 2017 Mar 21. PMID 29580594
- [Result] Cho EA, Kim KH, Park JY. [Effects of frozen gauze with normal saline and ice on thirst and oral condition of laparoscopic cholecystectomy patients: pilot study]. J Korean Acad Nurs. 2010 Oct;40(5):714-23. doi: 10.4040/jkan.2010.40.5.714. Korean. PMID 21157173